CLINICAL TRIAL: NCT02402504
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 1 - Acute Effects of Pulse Ingredients in Snack Products on Appetite, Blood Glucose, and Food Intake in Adults - Study 1
Brief Title: PERFECT Project - Part 1 - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:114-1
Record Dates: First submitted 2014-12-20; First posted 2015-03-30 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Extruded snack control (Placebo Comparator): 100% corn flour
  Interventions: Other: Control
- Extruded snack with small particle size pea flour (Experimental): 60% corn flour and 40% small particle size pea flour
  Interventions: Other: Small particle size pea flour
- Extruded snack with large particle size pea flour (Experimental): 60% corn flour and 40% large particle size pea flour
  Interventions: Other: Large particle size pea flour
- Extruded snack with lentil flour (Experimental): 60% corn flour and 40% lentil flour
  Interventions: Other: Lentil flour
- Extruded snack navy bean flour (Experimental): 60% corn flour and 40% navy bean flour
  Interventions: Other: Navy bean flour
- Extruded snack with pinto bean flour (Experimental): 60% corn flour and 40% pinto bean flour
  Interventions: Other: Pinto bean flour

INTERVENTIONS:
Other: Control — Non pulse extruded snack
  Arms: Extruded snack control
Other: Small particle size pea flour — Pulse extruded snack
  Arms: Extruded snack with small particle size pea flour
Other: Large particle size pea flour — Pulse extruded snack
  Arms: Extruded snack with large particle size pea flour
Other: Lentil flour — Pulse extruded snack
  Arms: Extruded snack with lentil flour
Other: Navy bean flour — Pulse extruded snack
  Arms: Extruded snack navy bean flour
Other: Pinto bean flour — Pulse extruded snack
  Arms: Extruded snack with pinto bean flour

SUMMARY:
The objectives are to test the acute effects of different extruded pulse snacks on: 1) post-prandial blood glucose, insulin and appetite for two hours, and 2) food intake two hours following consumption of pulse products.

The investigators hypothesize that snack products containing pulse ingredients will lead to lower blood glucose, insulin, appetite and food intake responses compared to non-pulse snack products.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year
* Competitive sports or athletic training at a high intensity
* Those unable to walk for an hour continuously

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0 - 200 min
  Measured in blood using intravenous catheter at 12 time points and used to calculate area under curve (AUC). Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits (Composite measure)
Food Intake | at 120 min
  Ad-libitum meal
Subjective Appetite | 0-200 min
  Measured by VAS questionnaire at 12 time points used to calculate area under curve (AUC) (Composite measure)

SECONDARY OUTCOMES:
Palatability of treatments | at 5 minutes
  Measured by VAS questionnaire
Palatability of meal | at 140 minutes
  Measured by VAS questionnaire
Energy and Fatigue | 0-200 min
  Measured by VAS questionnaire at 12 time points and use to calculate AUC. (Composite measure)
Physical Comfort | 0-200 min
  Measured by VAS questionnaire at 12 time points used to calculate area under curve (AUC). (Composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Johnston AJ, Mollard RC, Dandeneau D, MacKay DS, Ames N, Curran J, Bouchard DR, Jones PJ. Acute effects of extruded pulse snacks on glycemic response, insulin, appetite, and food intake in healthy young adults in a double blind, randomized, crossover trial. Appl Physiol Nutr Metab. 2021 Jul;46(7):704-710. doi: 10.1139/apnm-2020-0572. Epub 2020 Dec 21. PMID 33347383